CLINICAL TRIAL: NCT04080310
Title: Efficacy and Safety of Combination Therapy of Moderate-intensity Statin and Ezetimibe Compared to High-intensity Statin: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Combination Therapy of Moderate-intensity Statin and Ezetimibe Compared to High-intensity Statin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Si-Hyuck Kang, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YMC033
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination therapy group (Active Comparator): The combination therapy group will receive a single-pill combination of rosuvastatin 10 mg and ezetimibe 10 mg once daily.
  Interventions: Drug: Efficacy and safety of combination therapy of moderate-intensity statin and ezetimibe compared to high-intensity statin
- intensive statin group (Other): The subjects in the intensive statin group will receive rosuvastatin 20 mg once daily.
  Interventions: Drug: Efficacy and safety of combination therapy of moderate-intensity statin and ezetimibe compared to high-intensity statin

INTERVENTIONS:
Drug: Efficacy and safety of combination therapy of moderate-intensity statin and ezetimibe compared to high-intensity statin — This study is a multicenter, randomized, open-label, parallel, phase IV trial. The study is planned to include 272 patients with clinical ASCVD requiring optimal statin therapy.
  After enrollment, subjects are randomized into two groups in a 1:1 manner. patients in combination therapy group(rosuvastation 10mg and ezetimibe 10mg daily) will be provided a fixed-dose single pill comibation and patients in the intensive statin group will receive rosuvastatin 20mg daily.

SUMMARY:
This study is a multicenter, randomized, open-label, parallel, phase IV trial.

The purpose of this study efficacy and safety of combination therapy of moderate-intensity statin and ezetimibe compared to high-intensity statin.

DETAILED DESCRIPTION:
The study is planned to include 272 patients with a clinical atherosclerotic cardiovascular disease requiring optimal statin therapy.

After enrollment, subjects are randomized into two groups in a 1:1 manner. The combination therapy group will receive a single-pill combination of rosuvastatin 10 mg and ezetimibe 10 mg once daily.

The subjects in the intensive statin group will receive rosuvastatin 20 mg once daily.

Subjects will visit at weeks 12 and 24 to identify medication adherence and clinical side effects.

The primary endpoint of this study is a % change of low-density lipoprotein cholesterol at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 19 and 75 years
2. Presence of atherosclerotic cardiovascular disease Coronary artery disease

   * History of acute coronary syndrome
   * Stable or unstable angina
   * History of coronary revascularization Stroke or TIA Peripheral arterial disease, history of peripheral arterial revascularization
3. Patients who have been taking lipid-lowering agents (statin or ezetimibe) for ≥4 weeks at the time of randomization
4. Patients who gave informed consent

Exclusion Criteria:

1. Patients who have used lipid-lowering agents other than statin or ezetimibe within the last 3 months
2. A serum triglyceride on fasting >400 mg/dL
3. A history of muscular symptoms or rhabdomyolysis due to the use of statin
4. Hypersensitivity to rosuvastatin or ezetimibe
5. Labeled contraindications to rosuvastatin or rosuvastatin Severe renal impairment (CrCl <30 mL/min by Cockcroft-Gault formula or estimated GFR <30 mL/min / 1.73 m2 by MDRD equation) ALT, AST ≥3 × ULN or active liver disease CPK ≥3 × ULN
6. Enrollment of other clinical trials within 30 days
7. Any other issues that the treating physician assumes ineligible for participation in the trial

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
% change of low-density lipoprotein cholesterol | at 12 weeks
  %change of LDL-C = (LDL-C at 12 weeks) - (LDL-C at baseline)/LDL-C at baseline * 100

SECONDARY OUTCOMES:
% change of serum cholesterol level | at 12 and 24 weeks
  total cholesterol, LDL, HDL cholesterol, triglyceride (mg/dL)
% change of high-sensitivity C-reactive protein | at 12 and 24 weeks
  hs-CRP(mg/dL)
% change of fasting glucose | at 12 and 24 weeks
  fasting plasma glucose(mg/dL)
% change of homeostatic model assessment for insulin resistance(HOMA-IR) | at 12 and 24 weeks
  HOMA-IR = glucose * insulin / 405(glucose mg/dL , insulin uIU/mL)
proportion of participant with statin-associated muscle symptoms | at 12 and 24 weeks
  occurrence of statin-associated muscle symptoms
proportion of participant with creatinine phosphokinase elevation | at 12 and 24 weeks
  proportion of CPK elevation ≥4 or ≥10 upper normal of limit
proportion of participant with liver function test abnormality | at 12 and 24 weeks
  proportion of AST/ALT elevation ≥4 or ≥10 upper normal of limit
proportion of participant with major adverse cardiovascular and cerebrovascular events(MACCE) | at 12 and 24 weeks
  MACCE defined as a composite of the followings : cardiovascular death, acute myocardial infarction, unstable angina, stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided